CLINICAL TRIAL: NCT05219305
Title: Autogenous Mineralized Dentin Graft Compared to Partial Demineralized Tooth Graft and to Freeze-Dried Bone Allograft in Dental Implant Placement
Brief Title: Implant Stability in Autogenous Mineralized and Demineralized Dentin Grafts
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14063
Record Dates: First submitted 2022-01-18; First posted 2022-02-02 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Edentulous Alveolar Ridge
Keywords: dental implant,; autogenous dentin graft; autograft; allograft; bone graft

STUDY DESIGN:
Intervention Model Description: All participants originate from previous study ""Alveolar Ridge Preservation with evenly distributed experimental groups of FDBA, Mineralized, and Partially Demineralized Dentin Grafts". They have already been assigned and treated with different types of bone grafts. They were assigned groups via a computer randomization program.
Who Masked: Participant, Care Provider
Masking Description: Investigator completed randomization program and delivered grafting material to patient/dentist at time of grafting. Patients and providers still blinded as to which group they were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Freeze-Dried Bone Allograft (Experimental): edentulous site grafted with FDBA in previous study.
  Interventions: Device: Dental Implant Placement
- Partially-demineralized tooth graft (Experimental): edentulous site grafted with partially-demineralized tooth graft in the previous study.
  Interventions: Device: Dental Implant Placement
- mineralized tooth graft (Experimental): edentulous site grafted with mineralized tooth graft in the previous study.
  Interventions: Device: Dental Implant Placement

INTERVENTIONS:
Device: Dental Implant Placement — Placement in an edentulous site that was previously bone grafted in the prior study.

SUMMARY:
The bone grafting materials currently used in dentistry are autografts, allografts, xenografts, and alloplastic grafts. Among these different types of bone graft materials, autografts are considered to have the most predictable results due to their properties of osteogenesis, osteoinduction, and osteoconduction. However, bone autografts are rarely used due to the high morbidity associated with harvesting the bone graft from the patient with a second surgical site. Because of the increased risk to the patient with autogenous bone grafts, the current standard of care is an allograft, which is a bone graft harvested from cadaver sources such as Freeze-Dried Bone Allograft (FDBA). While allografts can only possess the qualities of osteoinduction and osteoconduction, they also have dramatically less morbidity due to the lack of a second surgical site.

Our null hypothesis states that: Experimental groups (mineralized, and partially demineralized dentin grafts) do not show positive changes in implant stability, survival, failure rate, probing pocket depth, and interproximal crestal bone level changes when compared to FDBA

Our alternative hypothesis states that: Experimental groups (mineralized, and partially demineralized dentin grafts) show similar or better results in terms of implant stability, survival, failure rate, probing pocket depth, and interproximal crestal bone level changes when compared to FDBA.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial that will assess the changes in implant stability, survival, failure rate, probing pocket depth, and interproximal crestal bone level changes recorded by ISQ (Implant Stability Quotient), probing pocket depths, x-ray, and direct clinical measurements which are routinely taken as a standard of care for the dental procedures of implant placement and evaluation. A non-invasive standardizing stent with a caliper will be used for direct measurements and for bitewing radiographs for the purpose of evaluating changes in bone level. Those measurements will be taken immediately at the time of implant placement, and 4-6 months after implant placement. Calibrated examiners will evaluate implant integration. This research will be carried out by a blinded examiner who will not know the grafted material type to prevent bias.

Interventions and follow-up appointments will be conducted at the University of Oklahoma (OU), Graduate Periodontics clinic. Approximately 5 visits are anticipated for each patient. Additional appointments may be needed depending on surgical complications that need attention or intervention. Following the completion of the study, the participants will be placed on appropriate recall schedules either at the Graduate Periodontics clinic or referred to their dentist of choice. The subject's information will not be used or distributed for future research studies even if identifiers are removed.

Patients from the previous study "Alveolar Ridge Preservation with evenly distributed experimental groups of FDBA, Mineralized, and Partially Demineralized Dentin Grafts". A total of 60 patients treated with Alveolar Ridge Preservation will be eligible for implant placement.

Protocol of the experiment is as follows:

1. Surgical intervention for implant placement (for all the groups).
2. 2-week follow-up after implant placement.
3. 6-week follow-up after implant placement.
4. 4-6 month follow-up after implant placement.
5. Restoration of the implant by the restorative dentist.
6. Data analysis

During the implant placement phase, at 4 to 6 months postoperative from the grafted sites, bone core sample will be collected using a trephine bur. Collection of sample with a trephine bur will come from area of bone being prepared for the dental implant and will be of a size that would have been removed during dental implant preparation anyway. This will occur during the same appointment as dental implant placement. The collected specimens will be labeled (name of the patient, date, and chart number) and sent to the OU Department of Oral Pathology where it will be analyzed for newly formed bone and the amount of residual bone graft material. This research will be carried out by a blinded examiner who will not know the grafted material type to prevent bias.

No population will be excluded based on race or gender. Patients under 18 years old will be excluded due to the ongoing growth potential of the alveolar bone at a younger age.

This study will be conducted at the University of Oklahoma, College of Dentistry, Department of Graduate Periodontics. Participants will be selected from patients of the College of Dentistry. Qualifying subjects will be scheduled for a screening examination appointment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years old. Current literature suggests that patients up to age 80 can safely receive dental implants. Patients older than 80 can get implant therapy with a rate of implant failure increase of 2.26%, but not statistically significant (Bertl et al. 2019)
* Well-controlled systemic disease.
* Able to understand and sign a written informed consent form and willing to fulfill all study requirements.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Currently smoking >10 cigarettes per day.
* History of head and/or neck radiotherapy in the past five years.
* Current use of bisphosphonates or history of IV bisphosphonate therapy.
* Pregnant, expecting to become pregnant, or lactating women.
* Presence of active periodontal disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Implant Stability as Measured with ISQ values of implant | 6 months
  Measurement of ISQ (Implant Stability Quotient) values of implant at follow-up appointments
Implant Failure Rate | 6 months
  Necessity of implant of implant removal from oral cavity
Probing pocket depth | 6 months
  measuring the depth of the periodontal pocket alongside the dental implant
Interproximal crestal bone level | 6 months
  radiographically assess bone level changes adjacent to dental implant

CONTACTS AND LOCATIONS:
Overall Officials: Robin Henderson, DDS, MS, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma College of Dentistry Graduate Periodontics, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No
Study records will be stored in a locked room and electronic records will be stored on an encrypted server, which meets the University IT Security requirements. Patient information will be kept within the University of Oklahoma.
  These records will be stored indefinitely on the server and available to copying and for future studies if requested under the supervision of a designated representative and in accordance with federal regulations.

REFERENCES:
- [Result] Jung RE, Fenner N, Hammerle CH, Zitzmann NU. Long-term outcome of implants placed with guided bone regeneration (GBR) using resorbable and non-resorbable membranes after 12-14 years. Clin Oral Implants Res. 2013 Oct;24(10):1065-73. doi: 10.1111/j.1600-0501.2012.02522.x. Epub 2012 Jun 15. PMID 22697628
- [Result] Murata, M. "Autogenous demineralized dentin matrix for maxillary sinus augmentation in human. The first clinical report." Journal of Dental Reseach., 82, B243.
- [Result] Ike M, Urist MR. Recycled dentin root matrix for a carrier of recombinant human bone morphogenetic protein. J Oral Implantol. 1998;24(3):124-32. doi: 10.1563/1548-1336(1998)0242.3.CO;2. PMID 9893518
- [Result] Saygin NE, Tokiyasu Y, Giannobile WV, Somerman MJ. Growth factors regulate expression of mineral associated genes in cementoblasts. J Periodontol. 2000 Oct;71(10):1591-600. doi: 10.1902/jop.2000.71.10.1591. PMID 11063392
- [Result] Emecen P, Akman AC, Hakki SS, Hakki EE, Demiralp B, Tozum TF, Nohutcu RM. ABM/P-15 modulates proliferation and mRNA synthesis of growth factors of periodontal ligament cells. Acta Odontol Scand. 2009;67(2):65-73. doi: 10.1080/00016350802555525. PMID 19031159
- [Result] Seo BM, Sonoyama W, Yamaza T, Coppe C, Kikuiri T, Akiyama K, Lee JS, Shi S. SHED repair critical-size calvarial defects in mice. Oral Dis. 2008 Jul;14(5):428-34. doi: 10.1111/j.1601-0825.2007.01396.x. PMID 18938268
- [Result] Kim YK, Kim SG, Byeon JH, Lee HJ, Um IU, Lim SC, Kim SY. Development of a novel bone grafting material using autogenous teeth. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Apr;109(4):496-503. doi: 10.1016/j.tripleo.2009.10.017. Epub 2010 Jan 8. PMID 20060336
- [Result] Kim YK, Kim SG, Yun PY, Yeo IS, Jin SC, Oh JS, Kim HJ, Yu SK, Lee SY, Kim JS, Um IW, Jeong MA, Kim GW. Autogenous teeth used for bone grafting: a comparison with traditional grafting materials. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Jan;117(1):e39-45. doi: 10.1016/j.oooo.2012.04.018. Epub 2012 Aug 30. PMID 22939321
- [Result] Koga T, Minamizato T, Kawai Y, Miura K, I T, Nakatani Y, Sumita Y, Asahina I. Bone Regeneration Using Dentin Matrix Depends on the Degree of Demineralization and Particle Size. PLoS One. 2016 Jan 21;11(1):e0147235. doi: 10.1371/journal.pone.0147235. eCollection 2016. PMID 26795024
- [Result] Binderman, Itzhak, Gideon Hallel, Casap Nardy, Avinoam Yaffe, and Lari Sapoznikov.
- [Result] Phillips DJ, Swenson DT, Johnson TM. Buccal bone thickness adjacent to virtual dental implants following guided bone regeneration. J Periodontol. 2019 Jun;90(6):595-607. doi: 10.1002/JPER.18-0304. Epub 2019 Jan 10. PMID 30578550
- [Result] Bertl K, Ebner M, Knibbe M, Pandis N, Kuchler U, Ulm C, Stavropoulos A. How old is old for implant therapy in terms of early implant losses? J Clin Periodontol. 2019 Dec;46(12):1282-1293. doi: 10.1111/jcpe.13199. Epub 2019 Nov 8. PMID 31529723
- [Result] Binderman, I., Hallel, G., Nardy, C., Yaffe, A., & Sapoznikov, L. (2014). A novel procedure to process extracted teeth for immediate grafting of autogenous dentin. J Interdiscipl Med Dent Sci, 2(154), 2.
- [Result] Korsch M. Tooth shell technique: A proof of concept with the use of autogenous dentin block grafts. Aust Dent J. 2021 Jun;66(2):159-168. doi: 10.1111/adj.12814. Epub 2021 Jan 25. PMID 33370452
- [Result] Howe MS, Keys W, Richards D. Long-term (10-year) dental implant survival: A systematic review and sensitivity meta-analysis. J Dent. 2019 May;84:9-21. doi: 10.1016/j.jdent.2019.03.008. Epub 2019 Mar 20. PMID 30904559